CLINICAL TRIAL: NCT03372928
Title: The Effects of Varying Essential Amino Acid Intakes on Resting and Post-exercise Skeletal Muscle and Whole-body Protein Kinetics During Negative Energy Balance
Brief Title: Essential Amino Acids and Protein Kinetics During Caloric Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: University of Arkansas (Other); Eastern Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-32HC
Record Dates: First submitted 2017-10-31; First posted 2017-12-14 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Muscle Protein Synthesis; Whole-body Protein Balance

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard EAA Dose (Experimental): EAA dose provided at 0.10 g/kg body mass
  Interventions: Dietary Supplement: Standard EAA
- High EAA Dose (Experimental): EAA dose provided at 0.30 g/kg body mass
  Interventions: Dietary Supplement: High EAA

INTERVENTIONS:
Dietary Supplement: Standard EAA — EAA provided relative to body mass at a standard dose (0.10 g/kg) during energy deprivation
  Arms: Standard EAA Dose
Dietary Supplement: High EAA — EAA provided relative to body mass at a high dose (0.30 g/kg) during energy deprivation
  Arms: High EAA Dose

SUMMARY:
The amount of essential amino acids (EAA) necessary to maximally stimulate muscle protein synthesis and optimize whole-body net protein balance during caloric deprivation has not been determined. This study will address that gap in knowledge by examining the resting and post-exercise muscle and whole-body protein kinetic responses to ingesting varying amounts of EAA after a 5 day period of negative energy balance. This study will provide the initial evidence to support the development of a recovery-based food product for military combat rations.

DETAILED DESCRIPTION:
Short-term negative energy balance downregulates muscle protein synthesis and upregulates whole-body proteolysis and amino acid (AA) oxidation, thereby increasing nitrogen excretion and exacerbating whole-body and skeletal muscle protein loss. Consumption of quality proteins high in essential amino acid (EAA) content may attenuate protein loss during energy deficit by restoring whole-body and skeletal muscle anabolic potential to that observed in a eucaloric state. During energy balance, muscle protein synthesis appears to be maximally stimulated after consuming 15 g of EAA at rest and after conventional resistance-type exercise. In response to a short-term energy deficit that downregulated basal muscle protein synthesis by as much as 27%, consuming 15 g (~7.5 g EAA) and 30 g (~15 g EAA) of whey protein after a bout of resistance exercise restored muscle protein synthesis rates to resting, fasted rates observed in the eucaloric state in a dose dependent manner. The effect of EAA intakes above 15 g on resting and post-exercise muscle protein synthesis and the whole-body protein anabolic response during acute energy deficit has not been determined. This study will assess resting and post-resistance exercise whole-body and skeletal muscle protein synthesis responses to across a spectrum of EAA intakes following a well-controlled, short-term (5-d) energy deficit (30% energy deficit). Using a randomized, double-blind, cross-over design, 20 resistance trained (≥ 2 d/wk for the past 6 mo) adults will undergo two, non-consecutive 5-d energy deficit periods, separated by a 14-d washout period. Resting and post-resistance exercise (single leg exercise model) whole-body protein turnover and skeletal muscle protein synthesis responses to two different doses of EAA (standard, 0.10 g/kg vs high, 0.30 g/kg) will be determined the morning after completing the 5-d energy deficit. This design will test the hypothesis that higher absolute doses of EAA are required to maintain resting and post-exercise anabolic responses during energy deficit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 35 years
* Body mass index < 30.0 kg/m2
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO)
* Resistance exercise trained defined by self-report as performing ≥ 2 sessions/wk for previous 6 mo
* Refrain from taking any nonsteroidal anti-inflammatory drugs (e.g., aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product for 10 days before starting and at least 5 days after completing the study
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes); vaping, chewing tobacco, caffeine, and dietary supplement use throughout the entire study period
* Supervisor approval for federal civilian employees and non-HRV active duty military personnel working within the US Army Natick Soldier Systems Center

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability as determined by the USARIEM Office of Medical Support and Oversight (OMSO)
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Abnormal PT/PTT test or problems with blood clotting
* History of complications with lidocaine
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Blood donation within 8-wk of beginning the study
* Pregnancy (self-report or results of urine pregnancy test before body composition testing)
* Unwillingness or inability to consume study diets or foods provided

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, PhD, Principal Investigator — Military Nutrition Division, USARIEM
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwin JA, Church DD, Hatch-McChesney A, Howard EE, Carrigan CT, Murphy NE, Wilson MA, Margolis LM, Carbone JW, Wolfe RR, Ferrando AA, Pasiakos SM. Effects of high versus standard essential amino acid intakes on whole-body protein turnover and mixed muscle protein synthesis during energy deficit: A randomized, crossover study. Clin Nutr. 2021 Mar;40(3):767-777. doi: 10.1016/j.clnu.2020.07.019. Epub 2020 Jul 22. PMID 32768315

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a cross-over design study. 19 volunteers completed both the standard and high EAA testing phases.
Groups:
- Low EAA First, Then High EAA: Participants received EAA provided relative to body mass at a standard dose (0.10 g/kg; LOW)) during energy deprivation first, then received EAA provided relative to body mass at a high dose (0.3 g/kg; HIGH) during energy deprivation.
- High EAA First, Then Low EAA: Participants received EAA provided relative to body mass at a high dose (0.30 g/kg; HIGH) during energy deprivation first, then received EAA provided relative to body mass at a low dose (0.1 g/kg; LOW) during energy deprivation.
Period: First Intervention (5 d Energy Deficit)
Arm/Group | Low EAA First, Then High EAA | High EAA First, Then Low EAA
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (14 d)
Arm/Group | Low EAA First, Then High EAA | High EAA First, Then Low EAA
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Period: Second Intervention (5 d Energy Deficit)
Arm/Group | Low EAA First, Then High EAA | High EAA First, Then Low EAA
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] | 25.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial, Resting Muscle Protein Synthesis Rates
Description: Assessed using stable isotope infusions of phenylalanine.
Time Frame: 3 hour measure of muscle protein synthesis
Measure: Mean (Standard Deviation); unit: percent per hour
Arm/Group | Standard EAA Dose | High EAA Dose
Number analyzed (Participants) | 19 | 19
percent per hour | 0.055 (0.01) | 0.061 (0.02)

2. Primary Outcome: Postprandial, Post-exercise Muscle Protein Synthesis Rates
Description: Assess using stable isotope infusions of phenylalanine.
Time Frame: 3 hour measure of muscle protein synthesis
Measure: Mean (Standard Deviation); unit: percent per hour
Groups:
- Standard EAA: Arm:
  EAA dose provided at 0.10 g/kg body mass
  Standard EAA: EAA provided relative to body mass at a standard dose (0.10 g/kg) during energy deprivation
- High EAA: Arm:
  EAA dose provided at 0.30 g/kg body mass
  High EAA: EAA provided relative to body mass at a high dose (0.30 g/kg) during energy deprivation
Arm/Group | Standard EAA | High EAA
Number analyzed (Participants) | 19 | 19
percent per hour | 0.055 (0.01) | 0.065 (0.02)

3. Primary Outcome: How Well Participants Suppress the Degradation of Body Proteins While Stimulating the Growth of New Proteins After Ingesting Varying Doses of EAA at Rest and After Exercise. Net Whole-body Protein Balance
Description: Assessed using stable isotope infusions of tyrosine. Net Whole-body Protein Balance is defined as whole-body protein synthesis - whole-body protein breakdown)
Time Frame: 3 hour measure of whole-body protein balance
Measure: Mean (Standard Deviation); unit: grams of protein per 180min
Groups:
- Standard EAA: Arm:
  EAA dose provided at 0.10 g/kg body mass
  Low EAA: EAA provided relative to body mass at a standard dose (0.10 g/kg) during energy deprivation
Arm/Group | Standard EAA | High EAA
Number analyzed (Participants) | 19 | 19
grams of protein per 180min | 2.7 (1.7) | 21.3 (3.4)

ADVERSE EVENTS:
Time Frame: 1 day
Description: non-serious adverse event
Groups:
- Low EAA First, Then High EAA: Low EAA Treatment: EAA dose provided at 0.10 g/kg body mass during first intervention, then EAA dose provided at 0.30 g/kg body mass during second intervention.
  Low EAA Treatment Period
- High EAA First, Then Low EAA: Low EAA Treatment: EAA dose provided at 0.30 g/kg body mass during first intervention, then EAA dose provided at 0.10 g/kg body mass during second intervention.
  Low EAA Treatment Period
- Low EAA First, Then High EAA: High EAA Treatment: EAA dose provided at 0.10 g/kg body mass during first intervention, then EAA dose provided at 0.30 g/kg body mass during second intervention.
  High EAA Treatment Period
- High EAA First, Then Low EAA: High EAA Treatment: EAA dose provided at 0.30 g/kg body mass during first intervention, then EAA dose provided at 0.10 g/kg body mass during second intervention.
  High EAA Treatment Period
Arm/Group | Low EAA First, Then High EAA: Low EAA Treatment | High EAA First, Then Low EAA: Low EAA Treatment | Low EAA First, Then High EAA: High EAA Treatment | High EAA First, Then Low EAA: High EAA Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low EAA First, Then High EAA: Low EAA Treatment (N=10) | High EAA First, Then Low EAA: Low EAA Treatment (N=10) | Low EAA First, Then High EAA: High EAA Treatment (N=10) | High EAA First, Then Low EAA: High EAA Treatment (N=10)
mild erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-serious adverse event, very mild erythema. No cellulitis or e/o abscess. No significant pain or tenderness. Diagnosis: contact dermitits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03372928/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03372928/ICF_001.pdf